CLINICAL TRIAL: NCT05668013
Title: A Phase 2b, Randomized, Double-Blind Long-Term Extension Study to Evaluate Pharmacokinetics, Efficacy, Safety, and Tolerability of TEV-48574 in Adult Patients With Moderate to Severe Ulcerative Colitis or Crohn's Disease Who Completed the Treatment Phase of the Dose-Ranging Study (RELIEVE UCCD LTE)
Brief Title: A Study to Evaluate the Long-Term Effect of TEV-48574 in Moderate to Severe Ulcerative Colitis or Crohn's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48574-IMM-20038; 2022-002593-89 (EudraCT Number); 2024-515027-11-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-12; First posted 2022-12-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Crohn Disease; Colitis, Ulcerative
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TEV-48574 Dose Regimen A for Ulcerative Colitis (UC) (Experimental): Administered by subcutaneous infusion for participants with UC
  Interventions: Drug: TEV-48574 Dose Regimen A
- TEV-48574 Dose Regimen A for Crohn's Disease (CD) (Experimental): Administered by subcutaneous infusion for participants with CD
  Interventions: Drug: TEV-48574 Dose Regimen A
- TEV-48574 Dose Regimen B for Ulcerative Colitis (UC) (Experimental): Administered by subcutaneous infusion for participants with UC
  Interventions: Drug: TEV-48574 Dose Regiment B
- TEV-48574 Dose Regimen B for Crohn's Disease (CD) (Experimental): Administered by subcutaneous infusion for participants with CD
  Interventions: Drug: TEV-48574 Dose Regiment B

INTERVENTIONS:
Drug: TEV-48574 Dose Regimen A — Subcutaneous (sc) administration using a commercial sc infusion system
  Other Names: duvakitug
  Arms: TEV-48574 Dose Regimen A for Crohn's Disease (CD); TEV-48574 Dose Regimen A for Ulcerative Colitis (UC)
Drug: TEV-48574 Dose Regiment B — Subcutaneous (sc) administration using a commercial sc infusion system
  Other Names: duvakitug
  Arms: TEV-48574 Dose Regimen B for Crohn's Disease (CD); TEV-48574 Dose Regimen B for Ulcerative Colitis (UC)

SUMMARY:
The primary objective of the study is to evaluate the efficacy of 2 different maintenance dose regimens of TEV-48574 subcutaneous (sc) administered every 4 weeks (Q4W) in adult participants with inflammatory bowel disease (IBD).

Secondary objectives of the study are to:

* evaluate the efficacy of 2 different maintenance dose regimens of TEV-48574 sc administered Q4W in adult participants with IBD
* evaluate the safety and tolerability of 2 different maintenance dose regimens of TEV-48574 sc administered Q4W in adult participants with IBD
* evaluate the immunogenicity of 2 different maintenance dose regimens of TEV-48574 sc administered Q4W in adult participants with IBD

The total duration for a participant in the double-blind period only is 66 weeks; and for a participant in the open-label extension (OLE) period, up to an additional 268 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance Period- Participants who achieved clinical response and/or clinical remission at week 14 of TV48574-IMM-20036 (the 14-week DRF study) or in the re-induction period of this study.
* Re-induction- Participants who did not achieve clinical response and/or clinical remission at week 14 of the TV48574-IMM-20036 DRF study

NOTE- Additional criteria may apply, please contact the investigator for more information

Exclusion Criteria:

* Participants who discontinued the TV48574-IMM-20036 study before scheduled week 14 visit (any reason including lack of efficacy, safety, or personal reasons)
* Participant has any concomitant conditions or treatments that could interfere with study conduct, influence the interpretation of study observations/results, or put the participant at increased risk during the study as judged by the investigator and/or the clinical study physician.
* Participant anticipates requiring major surgery during this study.
* Participant is currently pregnant or lactating or is planning to become pregnant or to lactate during the study or for at least 50 days after administration of the last dose of IMP in case of early termination. Any woman becoming pregnant during the study will be withdrawn from the study.

NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2031-03-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with moderate to severe ulcerative colitis (UC) who show clinical remission as defined by the Mayo score | Week 44
  Clinical remission based on modified (9-point rectal bleeding, stool frequency, and endoscopy) Mayo score of ≤2 points, which is defined by:
  * stool frequency subscore of 0 or 1,
  * rectal bleeding subscore of 0, and
  * endoscopic subscore of 0 or 1, where a score of 1 does not include "friability"
Number of participants with moderate to severe Crohn's disease (CD) who show an endoscopic response as defined by the Endoscopic Score for Crohn's Disease | Week 44
  Endoscopic response, defined as a decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) of at least 50% from DRF study baseline at week 44 in participants with CD

SECONDARY OUTCOMES:
Number of participants with moderate to severe UC with a clinical response as defined by Mayo score | Week 44
  Clinical response at week 44, defined as a decrease from baseline in the modified (9-point rectal bleeding, stool frequency, and endoscopy) Mayo score of at least 2 points AND at least a 30% reduction from DRF baseline with either a decrease in rectal bleeding subscore of at least 1 or an absolute rectal bleeding subscore of less than or equal to 1
Number of participants with moderate to severe UC with Endoscopic improvement as defined by Mayo score | Week 44
  Endoscopic improvement defined as a Mayo endoscopic subscore of 0 or 1
Number of participants with moderate to severe UC in Endoscopic remission as defined by Mayo score | Week 44
  Endoscopic remission defined as a Mayo endoscopic subscore of 0
Number of participants with moderate to severe UC with Corticosteroid-free clinical remission based on the modified Mayo score | Week 44
  Defined by clinical remission and corticosteroid-free for ≥12 weeks preceding week 44
Number of participants with moderate to severe CD with a clinical response based on Crohn's Disease Activity Index | Week 44
  Clinical response defined as a ≥100-point decrease from DRF baseline Crohn's Disease Activity Index (CDAI) score
Number of participants with moderate to severe CD in clinical remission as defined by CDAI score | Week 44
  Clinical remission defined as a CDAI score less than 150
Number of participants with moderate to severe CD with Corticosteroid-free endoscopic response based on SES-CD | Week 44
  Defined by endoscopic response and corticosteroid-free for ≥12 weeks preceding week 44
Number of participants with moderate to severe CD with Corticosteroid-free clinical remission based on CDAI | Week 44
  Defined by a CDAI score of <150 points and corticosteroid-free for ≥12 weeks preceding week 44
Number of participants who experience adverse events in the double-blind period | Up to Week 48
  Adverse events can include any of the following clinically significant changes in clinical laboratory test results (serum chemistry, hematology, and urinalysis), vital signs measurements (blood pressure, pulse rate, body temperature, and respiratory rate), 12-lead electrocardiogram (ECG), and injection site reactions.
Number of participants who experience adverse events in the open-label (OL) period | Up to 5 years after start of OL period
  Adverse events can include any of the following clinically significant changes in clinical laboratory test results (serum chemistry, hematology, and urinalysis), vital signs measurements (blood pressure, pulse rate, body temperature, and respiratory rate), 12-lead electrocardiogram (ECG), and injection site reactions.
Number of participants who stopped taking the investigational medicinal product (IMP) due to adverse events in the double-blind period | Up to Week 48
Number of participants who stopped taking the investigational medicinal product (IMP) due to adverse events in the open-label (OL) period | Up to 5 years after start of OL period
Number of participants with treatment emergent Anti-Drug Antibodies (ADA) | Weeks 0, 4, 8, 16, 28, 44, and 48
Number of ADA positive participants with the presence of neutralizing ADA | Weeks 0, 4, 8, 16, 28, 44, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D LLC
Locations (93):
- United States (18):
  - Teva Investigational Site 15556, San Diego, California
  - Teva Investigational Site 15357, Kissimmee, Florida
  - Teva Investigational Site 15375, Orlando, Florida
  - Teva Investigational Site 15359, Pinellas Park, Florida
  - Teva Investigational Site 15567, Gurnee, Illinois
  - Teva Investigational Site 15574, New Albany, Indiana
  - Teva Investigational Site 15367, Kansas City, Kansas
  - Teva Investigational Site 15575, Louisville, Kentucky
  - Teva Investigational Site 15358, Liberty, Missouri
  - Teva Investigational Site 15373, St Louis, Missouri
  - Teva Investigational Site 15369, Las Vegas, Nevada
  - Teva Investigational Site 15750, Beavercreek, Ohio
  - Teva Investigational Site 15559, Harlingen, Texas
  - Teva Investigational Site 15366, Katy, Texas
  - Teva Investigational Site 15374, San Antonio, Texas
  - Teva Investigational Site 15565, Southlake, Texas
  - Teva Investigational Site 15361, Tyler, Texas
  - Teva Investigational Site 15364, Salt Lake City, Utah
- Teva Investigational Site 33056, Vienna, Austria
- Bulgaria (3):
  - Teva Investigational Site 59243, Gorna Oryahovitsa
  - Teva Investigational Site 59197, Sofia
  - Teva Investigational Site 59196, Sofia
- Czechia (3):
  - Teva Investigational Site 54221, Brno
  - Teva Investigational Site 54222, Klatovy
  - Teva Investigational Site 54220, Slaný
- Georgia (2):
  - Teva Investigational Site 81052, Tbilisi
  - Teva Investigational Site 81053, Tbilisi
- Germany (4):
  - Teva Investigational Site 32793, Kiel
  - Teva Investigational Site 32795, Tübingen
  - Teva Investigational Site 32794, Ulm
  - Teva Investigational Site 32874, Wipperfürth
- Hungary (3):
  - Teva Investigational Site 51334, Budapest
  - Teva Investigational Site 51335, Budapest
  - Teva Investigational Site 51338, Vác
- Israel (2):
  - Teva Investigational Site 80179, Afula
  - Teva Investigational Site 80191, Beersheba
- Italy (3):
  - Teva Investigational Site 30285, Milan
  - Teva Investigational Site 30286, Milan
  - Teva Investigational Site 30284, Rozzano
- Japan (5):
  - Teva Investigational Site 84110, Kashiwa
  - Teva Investigational Site 84117, Minato
  - Teva Investigational Site 84114, Sakura
  - Teva Investigational Site 84116, Shinjuku
  - Teva Investigational Site 84111, Toyama
- Teva Investigational Site 41015, Lorenskog, Norway
- Poland (31):
  - Teva Investigational Site 53565, Bydgoszcz
  - Teva Investigational Site 53542, Częstochowa
  - Teva Investigational Site 53543, Elblag
  - Teva Investigational Site 53544, Gdansk
  - Teva Investigational Site 53546, Katowice
  - Teva Investigational Site 53560, Krakow
  - Teva Investigational Site 53548, Krakow
  - Teva Investigational Site 53512, Krakow
  - Teva Investigational Site 53547, Kłodzko
  - Teva Investigational Site 53515, Lodz
  - Teva Investigational Site 53518, Nowy Targ
  - Teva Investigational Site 53549, Poznan
  - Teva Investigational Site 53563, Poznan
  - Teva Investigational Site 53516, Poznan
  - Teva Investigational Site 53566, Poznan
  - Teva Investigational Site 53550, Sopot
  - Teva Investigational Site 53551, Staszów
  - Teva Investigational Site 53508, Szczecin
  - Teva Investigational Site 53519, Szczecin
  - Teva Investigational Site 53553, Torun
  - Teva Investigational Site 53554, Wadowice
  - Teva Investigational Site 53557, Warsaw
  - Teva Investigational Site 53570, Warsaw
  - Teva Investigational Site 53556, Warsaw
  - Teva Investigational Site 53555, Warsaw
  - Teva Investigational Site 53510, Wroclaw
  - Teva Investigational Site 53567, Wroclaw
  - Teva Investigational Site 53562, Wroclaw
  - Teva Investigational Site 53520, Wroclaw
  - Teva Investigational Site 53509, Zamość
  - Teva Investigational Site 53511, Łęczna
- Slovakia (5):
  - Teva Investigational Site 62074, Bardejov
  - Teva Investigational Site 62073, Bratislava
  - Teva Investigational Site 62071, Košice
  - Teva Investigational Site 62076, Prešov
  - Teva Investigational Site 62097, Prešov
- Spain (3):
  - Teva Investigational Site 31293, Huelva
  - Teva Investigational Site 31318, Santiago de Compostela
  - Teva Investigational Site 31292, Valencia
- Ukraine (8):
  - Teva Investigational Site 58327, Chernivtsi
  - Teva Investigational Site 58324, Ivano-Frankivsk
  - Teva Investigational Site 58329, Lviv
  - Teva Investigational Site 58325, Lviv
  - Teva Investigational Site 58332, Lviv
  - Teva Investigational Site 58322, Uzhhorod
  - Teva Investigational Site 58330, Vinnytsia
  - Teva Investigational Site 58331, Vinnytsia
- Teva Investigational Site 34305, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.